CLINICAL TRIAL: NCT00368810
Title: Response to Plasmodium Falciparum-Derived TLR Ligands in Severe and Uncomplicated Malaria in Mali
Brief Title: Study of Factors Involved in Resistance to Severe Malaria
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906104; 06-I-N104
Record Dates: First submitted 2006-08-22; First posted 2006-08-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-11-30

CONDITIONS: Malaria
Keywords: Children; Cross-Sectional; Glycosylphosphatidylinositol; Cytokines; Peripheral Blood Mononuclear Cells; Malaria
MeSH Terms: conditions — Malaria

SUMMARY:
This study will examine whether resistance to severe malaria is associated with weakening of a specific immune response (TLR-mediated pro-inflammatory cytokine response). Some children with mild malaria go on to develop severe disease, while others do not. The study will analyze certain substances in the blood to try to determine what factors may protect against severe malaria.

Healthy children and children 3 - 10 years of age with severe malaria who are being treated at l'H pital Gabriel Toure in Mamako, Mali, West Africa, may be eligible for this study. Participants have a mall sample of blood drawn from a vein and from two finger pricks.

DETAILED DESCRIPTION:
Malaria remains an important public health threat, responsible for over two million deaths annually, the majority among African children. The mechanisms underlying resistance to the most severe manifestations of malaria remain elusive. Severe malaria has been associated with high levels of pro-inflammatory cytokines that may contribute to the pathogenesis of cerebral malaria, severe anemia and acidosis. This response is thought to be driven primarily by glycosylphosphatidylinositol (GPI) anchors derived from erythrocyte-stage Plasmodium falciparum. It has been suggested that antibodies against GPI are responsible for resistance to severe malaria, which has led to efforts to develop a GPI-based vaccine. An alternative explanation for the development of resistance to severe malaria is down regulation of the innate pro-inflammatory response by repeated ligation of toll-like receptors (TLR) by GPI, or other putative P. falciparum-derived TLR ligands, such as hemozoin. This cross-sectional study at l'Hopital Gabriel Toure in Bamako, Mali, proposes to test the hypothesis that resistance to severe malaria is associated with an attenuation of the TLR-mediated pro-inflammatory cytokine response. After informed consent is obtained from the participant's parent or guardian, 2-3 mL of venous blood will be drawn from each of 60 children: 40 children presenting with acute P. falciparum infection (20 severe and 20 uncomplicated) and 20 healthy, P. falciparum uninfected controls. The blood will be tested for antibody titers against GPI and Merozoite Surface Protein-1 (MSP-1). Peripheral blood mononuclear cells (PBMCs) will be isolated and cultured with GPI, hemozoin, lipoteichoic acid (LTA), lipopolysaccharide (LPS), and cytosine-guanine dinucleotide (CpG). At 24 hours, supernatant will be collected and the following cytokines measured: IL-1, IL-6, IL-8, IL-10, IL-12, and TNF-alpha. A clearer understanding of the responsiveness to TLR ligands in children from malaria endemic areas may provide information on potential intervention strategies such as GPI-based vaccines or the use of TLR agonists as vaccine adjuvants.

ELIGIBILITY:
* INCLUSION CRITERIA -MALARIA PATIENTS:

  1. Males or females ages 3 to 10.
  2. Severe malaria as defined by positive blood smear for P. falciparum and need for hospitalization in accordance with the WHO definition of severe malaria (group I), or mild malaria as defined by positive blood smear for P. falciparum and triage to outpatient treatment (group II).
  3. Willingness of parent or guardian to have his or her child participate in the study as evidenced by the completed informed consent document.

INCLUSION CRITERIA -HEALTHY VOLUNTEERS:

1. Males or females ages 3 to 10.
2. No clinical evidence of malaria and negative blood smear.
3. No acute febrile or systemic illness.
4. Willingness of parent or guardian to have his or her child participate in the study as evidenced by the completed informed consent document.

EXCLUSION CRITERIA-MALARIA PATIENTS:

1. Active bleeding or hematocrit less than or equal to 15%.
2. Participation in a vaccine or drug trial within 30 days of starting this study.
3. Use of corticosteroids or immunosuppressive drugs within 30 days of starting this study.
4. Receipt of a live vaccine within past 4 weeks or killed vaccine within past 2 weeks prior to entry into the study.
5. Known history of HIV infection.

EXCLUSION CRITERIA-HEALTHY VOLUNTEERS:

1. Positive malaria smear.
2. Sibling of malaria patient.
3. Active bleeding or hematocrit less than or equal to 15%.
4. Participation in a vaccine or drug trial within 30 days of starting this study.
5. Use of corticosteroids or immunosuppressive drugs within 30 days of starting this study.
6. Receipt of a live vaccine within past 4 weeks or killed vaccine within past 2 weeks prior to entry into the study.
7. Known history of HIV infection.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120
Dates: Start 2006-02-21; Study Completion 2006-11-30

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Boutlis CS, Gowda DC, Naik RS, Maguire GP, Mgone CS, Bockarie MJ, Lagog M, Ibam E, Lorry K, Anstey NM. Antibodies to Plasmodium falciparum glycosylphosphatidylinositols: inverse association with tolerance of parasitemia in Papua New Guinean children and adults. Infect Immun. 2002 Sep;70(9):5052-7. doi: 10.1128/IAI.70.9.5052-5057.2002. PMID 12183552